CLINICAL TRIAL: NCT04477655
Title: Prone Positioning in Non-intubated Patients With Severe COVID-19: a Randomized Controlled Trial
Brief Title: Prone Positioning in Non-intubated Patients With COVID-19 Associated Acute Respiratory Failure
Acronym: PRO-CARF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Miguel Á Ibarra-Estrada, Principal investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 048/20
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: COVID-19; Severe; Prone positioning; High-flow nasal cannula
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard oxygen therapy (Active Comparator): Oxygen therapy through high flow nasal cannula (HFNC). Continuous monitoring of vital signs. Inspired fraction of oxygen will be titrated to maintain a capillary saturation of ≥92%. Prone positioning will be allowed as a rescue therapy.
  Interventions: Procedure: Standard oxygen therapy
- Awake prone positioning (Experimental): Oxygen therapy through high flow nasal cannula (HFNC). Patients will be asked to remain in prone position throughout the day as long as possible, with breaks according to tolerance. Pillows will be offered for maximizing comfort at chest, pelvis and knees. Monitoring of vital signs will not be suspended. Inspired fraction of oxygen will be titrated to maintain a capillary saturation of ≥92%.
  Interventions: Procedure: Awake prone positioning

INTERVENTIONS:
Procedure: Awake prone positioning — Patients will be asked to remain in prone position or lateral decubitus throughout the day as long as possible.
  Arms: Awake prone positioning
Procedure: Standard oxygen therapy — Oxygen therapy through high flow nasal cannula (HFNC). Inspired fraction of oxygen will be titrated to maintain a capillary saturation of ≥92%
  Arms: Standard oxygen therapy

SUMMARY:
Besides protective ventilation with low tidal volumes, prone positioning is a proven intervention to decrease mortality in mechanically ventilated patients with moderate-severe acute respiratory distress syndrome. However, the evidence of this strategy in awake non-intubated patients is scarce. The investigators will perform a randomized controlled trial to define if prone positioning can reduce the requirement of mechanical ventilation.

DETAILED DESCRIPTION:
Despite ongoing trials of antivirals and immunomodulatory therapies against COVID-19, the treatment of moderate/severe disease is mainly supportive, including oxygen therapy and invasive mechanical ventilation when impending respiratory failure is established. Moreover, the associated mortality among mechanically intubated patients is overwhelmingly high. Prone position relieves the dependent lung regions from the compressive forces of the mediastinum's weight, leading to homogenization of the gas:tissue ratio between ventral and dorsal lung regions. According to a few case series, and observational non-randomized studies with small sample sizes, there is a consistent improvement in oxygenation in COVID-19 patients during prone positioning, however there are no clinical evidence that this improvement is associated with a decrease in the risk of invasive mechanical ventilation. Considering that prone positioning is a low cost, low risk and widely available therapy, more high quality evidence is needed, to determine if the benefits of prone positioning in awake patients also include a lower requirement of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed COVID-19, and requirement of a fraction of inspired oxygen (FiO2) ≥30% through high-flow nasal cannula (HFNC) to maintain a capillary saturation of ≥90%

Exclusion Criteria:

* Less than 18 years-old
* Pregnancy
* Patients with immediate need of invasive mechanical ventilation
* Contraindications for prone positioning therapy
* Do-not-resuscitate or do-not-intubate order
* Refusal of the patient or decision maker to enroll in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Intubation rate | 28 days

SECONDARY OUTCOMES:
Total hours of prone position at day | 28 days
Total number of prone sessions at day | 28 days
Hours of the longest prone session each day | 28 days
Change in oxygenation 1-hour after first prone session | 1 hour
Change in the ROX-index 1-hour after first prone session | 1 hour
  The change in the Ratio of Oxygen saturation to respiratory rate (ROX-index)
Total days of prone positioning therapy | 28 days
Adverse effects of prone positioning therapy | 28 days
Mechanical ventilation days | 28 days
Intensive care unit length of stay | 28 days
Hospital length of stay | 28 days
Hospital mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ibarra-Estrada, Principal Investigator — Investigator
Locations (2):
- Mexico (2):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Hospital General de Occidente, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibarra-Estrada M, Li J, Pavlov I, Perez Y, Roca O, Tavernier E, McNicholas B, Vines D, Marin-Rosales M, Vargas-Obieta A, Garcia-Salcido R, Aguirre-Diaz SA, Lopez-Pulgarin JA, Chavez-Pena Q, Mijangos-Mendez JC, Aguirre-Avalos G, Ehrmann S, Laffey JG. Factors for success of awake prone positioning in patients with COVID-19-induced acute hypoxemic respiratory failure: analysis of a randomized controlled trial. Crit Care. 2022 Mar 28;26(1):84. doi: 10.1186/s13054-022-03950-0. PMID 35346319
- [Derived] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Derived] Ibarra-Estrada MA, Marin-Rosales M, Garcia-Salcido R, Aguirre-Diaz SA, Vargas-Obieta A, Chavez-Pena Q, Lopez-Pulgarin JA, Mijangos-Mendez JC, Aguirre-Avalos G. Prone positioning in non-intubated patients with COVID-19 associated acute respiratory failure, the PRO-CARF trial: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 23;21(1):940. doi: 10.1186/s13063-020-04882-2. PMID 33225990